CLINICAL TRIAL: NCT01581697
Title: Impact of Consumption of Oats in Lipid Profile of Children and Adolescents With Dyslipidemia at the Outpatient Clinic of Reference in Preventive Pediatric Cardiology at the Institute of Cardiology of Rio Grande do Sul
Brief Title: Impact of Consumption of Oats in Lipid Profile of Children and Adolescents With Dyslipidemia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Collaborators: Quaker Oats Company (Industry); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Impacto do consumo de aveia no perfil lipídico de crianças e adolescentes com dislipidemia atendidas no ambulatório de referência em cardiologia pediátrica preventiva do instituto de cardiologia do rio grande do sul, Institute fo Cardiology of Rio Grande do Sul
Other Study IDs: up 4100/07
Record Dates: First submitted 2012-04-17; First posted 2012-04-20 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Atherosclerosis; Hypercholesterolemia
Keywords: oat; cholesterol; children; adolescent; Level reduction of ceric cholesterol
MeSH Terms: conditions — Atherosclerosis; Hypercholesterolemia; Gyrate Atrophy

ARMS (1):
- Oat bran (Experimental)
  Interventions: Dietary Supplement: Oat bran

INTERVENTIONS:
Dietary Supplement: Oat bran

SUMMARY:
Atherosclerosis is the leading cause of death and disability in adults. However, investigations suggest that the basic pathology of heart disease as more severe myocardial infarction which usually reach mainly middle-aged or above, starts from childhood. Hypercholesterolemia is one of the most important risk factors for atherosclerosis in adults and children, is associated with early deposition of lipids in the aorta and coronary arteries.

Among other recommendations for prevention and treatment of heart disease and risk factors, is the recommendation to encourage the intake of soluble fiber. The oats, a major source of soluble fiber, has been recognized as a potential component of the diet to lower blood cholesterol levels, this effect is attributed mainly to the beta-glucan, a type of soluble fiber present in large quantities in oats. In 1997 the Food and Drug Administration admitted that the oat bran, oat flakes and oatmeal may have beneficial effects for health with the recommendation of daily intake of 3g of beta-glucan from oats and a food that brings a claim for promotion health, must provide, without enrichment, at least 1 gram of beta-glucan per serving.

The objective of this project will be compared by randomized clinical trial, the impact of intake of oats, for 8 weeks in the lipid profile of children and adolescents with dyslipidemia.

Will be included in the study 120 volunteers aged between 5 and 16 years who are in nutritional monitoring for at least 1 month. The subjects will be randomly divided into 2 groups, with a control group and another intervention will receive 3 tablespoons of soup filled with oat bran, which corresponds to 3g of beta-glucan, along with breakfast, lunch and dinner. Patients will be monitored with consultations on the 2nd, 4th and 8th weeks of treatment. Blood sample will be performed, to obtain the lipid profile of patients, at the beginning and end of the study. To compare the groups are used Student's t and squared chi. The alpha of 0.05 is considered critical. The program will be used Statistical Package for the Social Sciences (SPSS) version 15.0.

It is expected a decrease in serum levels of total cholesterol and LDL-c. Thus, living habits and healthy alternatives to prevent these risk factors should be done since childhood, especially in children who already have cholesterol levels of change.

ELIGIBILITY:
Inclusion Criteria:

* Male/Female
* Age limits 5 years-16 years

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Cardiologia do Rio Grande do Sul - Fundação Universitária de Cardiologia, Porto Alegre, Rio Grande do Sul, Brazil